CLINICAL TRIAL: NCT03696290
Title: A Trial of the Safety, Tolerability and Efficacy of 2 Doses of Cayston (Aztreonam Lysine) Compared to Placebo in Participants With Bronchiectasis
Brief Title: Value of Inhaled Treatment With Aztreonam Lysine in Bronchiectasis
Acronym: VitalBE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: University of Dundee (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, James Chalmers, Professor, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016RC27; 2018-001590-24 (EudraCT Number)
Record Dates: First submitted 2018-09-07; First posted 2018-10-04 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Bronchiectasis Adult
Keywords: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Aztreonam

STUDY DESIGN:
Intervention Model Description: Multi-centre randomised double-blind placebo controlled parallel group trial with four treatment arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Trail management team will also be masked. A bespoke online randomisation system will be used to generate the treatment codes for each participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Aztreonam lysine, 3 doses per day (Active Comparator): 3 doses per day of nebulised Aztreonam lysine (75 mg) for 1 month, followed by 1 month off treatment. The month on, month off regimen will be repeated for a total peroid of 12 months.
  Interventions: Drug: Aztreonam lysine
- Placebo, 3 doses per day (Placebo Comparator): 3 doses per day of nebulised placebo (5 mg lactose monohydrate) for 1 month, followed by 1 month off treatment. The month on, month off regimen will be repeated for a total peroid of 12 months.
  Interventions: Other: Placebo
- Aztreonam lysine, 2 doses per day (Active Comparator): 2 doses per day of nebulised Aztreonam lysine (75 mg) for 1 month, followed by 1 month off treatment. The month on, month off regimen will be repeated for a total peroid of 12 months.
  Interventions: Drug: Aztreonam lysine
- Placebo, 2 doses per day (Placebo Comparator): 2 doses per day of nebulised placebo (5 mg lactose monohydrate) for 1 month, followed by 1 month off treatment. The month on, month off regimen will be repeated for a total peroid of 12 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aztreonam lysine — Nebulised aztreonam lysine 75mg
  Other Names: Cayston
  Arms: Aztreonam lysine, 2 doses per day; Aztreonam lysine, 3 doses per day
Other: Placebo — Nebulised lactose monohydrate 5mg
  Other Names: Lactose monohydrate
  Arms: Placebo, 2 doses per day; Placebo, 3 doses per day

SUMMARY:
A randomised controlled trial of the safety, tolerability and effectiveness of Cayston Cayston (Aztreonam Lysine) compared to placebo in participants with bronchiectasis.

Bronchiectasis not due to cystic fibrosis is a chronic inflammatory disease characterised by cough, sputum production and frequent respiratory tract infections. There are currently no licensed therapies for bronchiectasis approved by regulators in the United States or Europe. The disease has a high morbidity, particularly in the presence of chronic P. aeruginosa and other chronic Gram-negative infections.

This trial will test the hypothesis that 12 months treatment with Aztreonam lysine for inhalation will be safe and well tolerated, and will result in a significant increase in the time to first pulmonary exacerbation in participants with bronchiectasis and a history of frequent exacerbations.

This is a multi-centre randomised double-blind placebo controlled parallel group trial with four treatment arms. It will enroll 100 bronchiectasis patients with a history of at least 3 exacerbations in the previous year and the presence of chronic Gram-negative infection in sputum at screening. Patients will be treated following a one month on, one month off treatment regimen for 12 months.

The primary objective is to evaluate the safety and tolerability of Aztrenam lysine in these patients by recording adverse events and trial treatment withdrawals.

DETAILED DESCRIPTION:
Chronic neutrophilic inflammation is a feature of bronchiectasis and the levels of neutrophilic inflammation predict the risk of future exacerbations. Neutrophilic inflammation is highest in participants with P. aeruginosa and other Gram negative pathogens and inflammation can be suppressed by inhaled antibiotic treatment . There is therefore a strong rationale for the effectiveness of inhaled antibiotic treatment in bronchiectasis.

Studies of inhaled antibiotics in bronchiectasis have given mixed results to date. Several open label studies in the late 1980's, testing nebulised β-lactams, demonstrated reduced sputum purulence, sputum volume and improvements in inflammatory markers. In an early phase II double-blind placebo-controlled trial by Barker et al. nebulised tobramycin significantly reduced the primary outcome of P. aeruginosa bacterial load but was poorly tolerated by some participants. Subsequently a single centre randomised controlled trial of nebulised gentamicin for 12 months reported significant benefits but was limited by open label design and small sample size. Haworth et al recruited 144 participants with chronic P. aeruginosa infection and randomized participants to nebulised colistin or placebo. The trial narrowly failed to meet its primary end-point (colistin group 165 days versus placebo 111 days; p=0.11). In the secondary end-points, a large improvement in quality of life using the SGRQ was noted (mean difference -10.5 points; p=0.006).

Aztreonam is an inhaled antibiotic licensed for treatment in cystic fibrosis. Two recent phase III trials in bronchiectasis randomised 266 (AIR-BX1) and 274 (AIR-BX2) participants to Aztreonam 75mg three times daily or placebo over the course of two 28-day treatment cycles (with 28 days off treatment between cycles). The primary outcome was the newly developed Quality of Life Bronchiectasis (QoL-B) questionnaire. Unfortunately the trial failed to meet its primary end-point, with a significant change observed in the QOL-B respiratory symptom score in AIR-BX2 but not in AIR-BX1. Treatment related adverse effects were also increased in the Aztreonam treated participants.

Likely explanations for the difficulties encountered in this previous trial include that the trial population was quite heterogeneous, with many participants having no history of exacerbations and appearing to have relatively mild disease. Many patients did not have a history exacerbations in this trial whereas the ERS bronchiectasis guidelines suggest limiting inhaled antibiotic use to patients with a history of 3 or more exacerbations per year. The characteristics of the included participants included high rates of pulmonary non-tuberculous mycobacterial disease and COPD. Nadig and Flume compared the characteristics of included participants in this trial to their own population of participants with severe bronchiectasis treated with inhaled antibiotics and identified little correlation, suggesting that the trials included a skewed population that was not representative of real-life clinical practice (Nadig and Flume AJRCCM 2016).

In addition, no dose finding studies were performed in bronchiectasis. The dose of 75mg three times daily was chosen based on efficacy and safety in cystic fibrosis. The rates of adverse events appear to be higher in bronchiectasis suggesting that doses selected for CF may not be fully appropriate for participants with non-CF bronchiectasis. Whether lower doses may have efficacy and better safety has not been investigated.

There is a need to determine the safety and efficacy of Aztreonam lysine in participants with bronchiectasis and a history of frequent exacerbations.

The researchers hypothesise that Aztreonam lysine will be safe and well tolerated and will reduce the frequency of exacerbations in participants with bronchiectasis and a history of frequent exacerbations. This trial will test two different doses of Aztreonam lysine compared to placebo. The efficacy and safety of Aztreonam is supported by the evidence for Aztreonam in cystic fibrosis where Aztreonam prolonged the time to first exacerbation by 21 days compared to placebo and improved quality of life. The AIR-BX studies evaluated Aztreonam for inhalation for only 2 treatment cycles. They showed suppression of chronic Gram-negative airway bacterial load but were not designed to evaluate the impact of Aztreonam on the frequency or time to first exacerbation. No attempt to identify the optimal dose was made. The incidence of treatment related adverse effects was increased in AIR-BX1 but was more balanced in AIR-BX2, a trial conducted primarily in European bronchiectasis participants. The reason for this imbalance is unknown.

The researchers hypothesise that 12 months treatment with Aztreonam lysine for inhalation will be safe and well tolerated, and will result in a significant increase in the time to first pulmonary exacerbation in participants with bronchiectasis and a history of frequent exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Able to give informed consent
* Clinical diagnosis of Bronchiectasis
* CT scan of the chest demonstrating bronchiectasis in 1 or more lobes
* A history of at least 3 exacerbations in the previous 12 months
* Bronchiectasis severity index score >4
* Pseudomonas aeruginosa or other Gram-negative respiratory pathogen detected in sputum or bronchoalveolar lavage on at least 1 occasion in the previous 12 months.
* A sputum sample that is culture positive for P. aeruginosa or other Gram-negative respiratory pathogens sent at the screening visit and within 28 days of randomization. Pre-specified eligible organisms include Eschericia coli, Haemophilus influenzae, Moraxella catarrhalis, Klebsiella pneumoniae, Proteus mirabilis, Serratia marcescens, Achromobacter, Enterobacter and Stenotrophomonas maltophilia

Exclusion Criteria:

* Participant has cystic fibrosis
* Immunodeficiency requiring replacement immunoglobulin.
* Active tuberculosis or nontuberculous mycobacterial infection (defined as currently under treatment, or requiring treatment in the opinion of the investigator).
* Recent significant haemoptysis (a volume requiring clinical intervention, within the previous 4 weeks).
* Treatment with inhaled, systemic or nebulized anti-Pseudomonal antibiotics in the 28 days prior to randomization
* Oral macrolides which have been taken for a period of less than 3 months prior to the start of the trial.
* Treatment of an exacerbation and receiving antibiotic treatment within 4 weeks of randomization
* Primary diagnosis of COPD associated with >20 pack years smoking history.
* History of poorly controlled asthma or a history of bronchospasm with inhaled antibiotics.
* Pregnant or lactating females.
* Participants with FEV1 <30% predicted value at screening.
* Previous history of intolerance to Aztreonam or bronchospasm reported with any other inhaled anti-bacterial.
* Glomerular filtration rate (eGFR) below 30ml/min/1.73m2 or requiring dialysis. This will be determined at screening.
* Use of any investigational drugs within five times of the elimination half-life after the last trial dose or within 30 days, whichever is longer.
* Unstable co-morbidities (cardiovascular disease, active malignancy) which in the opinion of the investigator would make participation in the trial not in the participants best interest.
* Long term oxygen therapy
* Women of child bearing age or male partners of women of child bearing age and not practicing a method of acceptable birth control (see below)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-10-19 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
The number of adverse events, serious adverse events and trial treatment withdrawals in order to evaluate the safety and tolerability of Aztreonam lysine | 12 months
  Adverse events, serious adverse events and trial treatment withdrawals will be recorded and a comparison made between the 4 treatment groups

SECONDARY OUTCOMES:
To determine the effect of Aztreonam Lysine on time to first protocol-defined pulmonary exacerbation | 12 months
  Time to first exacerbation, measured in days
To determine the effect of Aztreonam lysine on the frequency of protocol-defined exacerbations over 12 months | 12 months
  Number of exacerbation events
To determine the effect of Aztreonam lysine on quality of life using the St Georges Respiratory questionnaire | 12 months
  St. Georges Respiratory Questionnaire is a 50-item questionnaire developed to measure health status (quality of life) in patients with diseases of airways obstruction.
  Scores are calculated for three domains:
  Symptoms, Activity and Impacts (Psycho-social) as well as a total score. The score correlates significantly with other measures of disease activity such as cough, dyspnoea, 6-min walk test and FEV1 as well as other measures of general health. http://www.healthstatus.sgul.ac.uk/sgrq
To determine the effect of Aztreonam lysine on quality of life using the Quality of Life (QOL) Bronchiectasis Questionnaire | 12 months
  QOL Bronchiectasis Questionnaire is a new, disease-specific health-related qualify of life (HRQOL) measure for adults with non-CF bronchiectasis. It has several different scales, including symptoms, physical, social and emotional functioning. It was developed using the FDA Guidance on Patient-Reported Outcomes1 beginning with interviews with health care providers, open-ended interviews with patients, item generation, cognitive testing and then a national psychometric validation. It is being used internationally in several clinical trials. It is also used clinically during routine clinic visits.
  Speight, J., & Barendse, S. M. (2010). FDA guidance on patient reported outcomes. BMJ, 340. The questionnaire measures functioning in a variety of domains, including Physical Functioning, Role Functioning, Vitality, Emotional Functioning, Social Functioning, Treatment Burden, Health Perceptions, and Respiratory Symptoms. High scores indicate better health-related quality of life.
To determine the effect of Aztreonam lysine on quality of life using the Bronchiectasis Health Questionnaire | 12 months
  The BHQ is a brief, valid and repeatable, self-completed health status questionnaire for bronchiectasis that generates a single total score. It can be used in the clinic to assess bronchiectasis from the patient's perspective.
  "The development and validation of the Bronchiectasis Health Questionnaire Arietta Spinou, Richard J. Siegert, Wei-jie Guan, Amit S. Patel, Harry R. Gosker, Kai K. Lee, Caroline Elston, Michael R. Loebinger, Robert Wilson, Rachel Garrod, Surinder S. Birring. European Respiratory Journal 2017 49: 1601532
To determine the effect of Aztreonam lysine on pulmonary function | 12 months
  Spirometry, specifically the forced expiratory volume in 1 minute
Bacterial load at the end of the first treatment cycle | 28 days
  Colony Forming Units per mililitre (CFU/ml)

OTHER OUTCOMES:
To determine the impact of Aztreonam lysine on the time to first exacerbation, including all clinically treated exacerbations | 12 months
  Time to first exacerbation (protocol defined and non-protocol defined)
To determine the compliance with medication regimes | 12 months
  Missed doses of medication will be counted for each treatment group

CONTACTS AND LOCATIONS:
Overall Officials: James Chalmers, MBChB, MRCP, Principal Investigator — University of Dundee
Locations (14):
- United Kingdom (14):
  - Torbay Hospital, Torquay, Devon
  - Royal Papworth hospital NHS Foundation Trust, Cambridge
  - Cardiff & Vale University Local Health Board, Cardiff
  - University Hospitals of Derby and Burton NHS Foundation Trust, Derby
  - NHS Tayside, Dundee
  - NHS Lanakrshire University Hospital Hairmyres, East Kilbride
  - The Princess Alexandra Hospital NHS Trust, Harlow
  - Liverpool Heart and Chest Hospital, Liverpool
  - Aintree University Hospital, Liverpool
  - Royal Brompton & Harefield NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust - Wythenshawe Hospital, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - University hospital Southampton NHS Foundation Trust, Southampton
  - NHS Lanarkshire: University Hospital Wishaw, Wishaw

IPD SHARING:
Plan to Share IPD: No